CLINICAL TRIAL: NCT04828668
Title: A Single-Blind, Randomized, Placebo Controlled, Study to Evaluate the Benefits and Safety of Endourage Targeted Wellness Formula C™ Sublingual Drops in People With Post -Acute COVID-19 Syndrome (PACS).
Brief Title: Study to Evaluate Benefits & Safety of Endourage Formula C™ Oral Drops in People With Post-Acute COVID-19 Syndrome.
Acronym: "BAC-PAC"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endourage, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ENDO-402-2021
Record Dates: First submitted 2021-03-10; First posted 2021-04-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A total of 60 (sixty) participants who meet inclusion and exclusion criteria will be randomized and enrolled in a 1:1 ratio of study product (Formula C) vs. placebo.
  Group 1: 30 participants will be randomized to masked active study product (Formula C) for 28-days; they will continue to the open label extension phase (with commercially available product for an additional 28-days when they will receive commercially available product.
  Group 2: 30 participants will be randomized to placebo for 28-days; they will roll-over to the open label extension phase of study product (Formula C) for an additional 28-days when they will receive commercially available product.
  At the completion of the treatment period, the participants will be followed for 14-days.
Who Masked: Participant
Masking Description: Treatment period 1 will utilize masked study product labels with subject ID. Treatment period 1 will utilized unmasked / open-label study product with subject ID.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formula C (Experimental): 30 participants will be randomized to masked active study product (Formula C) for 28-days; they will continue to the open label extension phase (with commercially available product for an additional 28-days when they will receive commercially available product.
  Interventions: Dietary Supplement: Targeted Wellness Formula C™ Sublingual Drops - 1200mg - 30 mL (Formula C)
- Placebo (Placebo Comparator): 30 participants will be randomized to placebo for 28-days; they will roll-over to the open label extension phase of study product (Formula C) for an additional 28-days when they will receive commercially available product.
  Interventions: Dietary Supplement: Targeted Wellness Formula C™ Sublingual Drops - 1200mg - 30 mL (Formula C)

INTERVENTIONS:
Dietary Supplement: Targeted Wellness Formula C™ Sublingual Drops - 1200mg - 30 mL (Formula C) — Hemp seed oil
  Other Names: Placebo

SUMMARY:
This study will explore the contribution of CBD oral drops in persons experiencing symptoms of Post Acute COVID Syndrome or "PACS".

DETAILED DESCRIPTION:
At present, conventional medical and rehabilitation therapies have not consistently been effective for people with PACS, and in fact some symptoms have been observed to worsen over time. This inconsistency in clinical response has created a need for alternative treatment options to be explored. CBD presents a novel approach that warrants further investigation.

After review and approval by an Institutional Review Board (IRB), potential study participants will be recruited from on-line support groups who have identified themselves as persons experiencing post-acute COVID-19 syndrome also known as (long-haulers syndrome).

The study will be registered on the www.clincaltrials.gov website and will accept referrals from targeted clinics who refer their patients to the investigational site listed and individuals can also self-refer to the study center team.

Subjects will be evaluated weekly using telemedicine procedures. At completion of study, there will be a 7-day and 14-day follow up telemedicine visit to assess for continued benefit and/or re-emergence of symptoms/relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older who can provide informed consent.
2. Persons who have been diagnosed with COVID-19 and now in post-acute recovery phase.
3. Persons who are in care with access to primary care for post COVID infection or PACS.
4. Ability to read and write in the English language and follow study-related procedures.
5. Ability to have mail/ study drug delivered to an address and/or P.O. Box in the recipient's name.
6. Ability to participate in telemedicine visits/communication.
7. If a woman of childbearing age, willing to use a dual method of contraception (barrier and/or hormonal).

Exclusion Criteria:

1. Active illicit or non-prescribed drug use.
2. Concomitant use of benzodiazepines.
3. Concomitant use of an immune suppressant agent, e.g., prednisone.
4. Documented history and active treatment for seizure disorder.
5. Transaminase elevation.
6. Active autoimmune disorder.
7. Hepatitis C infection (currently on therapy and/or any transaminitis elevation).
8. Hepatitis B infection (currently on therapy and/or any transaminitis elevation).
9. Human Immune Deficiency Virus (HIV-1 or HIV-2) infection that is newly diagnosed or untreated.
10. Any form of mental impairment that will/could hinder safe participation in the study.
11. Pregnancy or breast-feeding.
12. Any condition that in the opinion of the investigator would be harmful or detrimental to the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Reduction in patient reported outcomes measures on the Patient Reported Outcomes Measurement Information System (PROMIS ®) assessment tools. | 56-days (designated time points)
  PROMIS® is a set of patient-centered instruments used to measure various patient reported outcomes.
  Measures are scored on the T-score metric of which 50 is the mean of a relevant baseline population with 10 being the standard deviation of that population.
  A score of 40 is one stndard deviation less than and a score of 60 is one standard deviation greater than the mean of the baseline or reference population.
  High scores suggest more of what is being measured (e.g., more fatigue, more shortness of breath) and a lower score suggest improvement in symptoms or complaints assessed depending on symptom or complaint being measured.
PATIENT GLOBAL IMPRESSION OF CHANGE (PGIC) | 56-days (designated time points)
  This scale evaluates various aspects of patients' health and assesses if there has been an improvement or decline in clinical status. Scale associated with subjective responses range 1-7 (from no change or a one through a great deal better and considerable improvement that has made all the difference or a seven), higher ratings indicate improved sympomtoms (responders) versus those reporting lower scores suggesting no change or a worsening of their condition (non-responders).

SECONDARY OUTCOMES:
Study product related adverse events and side effects. | 56-days (designated time points)
  Daily diary entries and clinical interview at scheduled visit; the number of participants with treatment related events as measured by grading scale of the Common Terminology Criteria for Adverse Events (CTCAE), grade 1-IV (one through four) and using descriptor terms, mild, moderate, severe. Additionally, any adverse event meeting serious adverse event criteria will be collected and reported. Frequency summary tables of all adverse events/serious adverse events will be tabulated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Young, PhD, NP, Principal Investigator — JOEL S ERICKSON, MD & THOMAS P YOUNG, PHD NP
Locations (1):
- Thomas P Young, Novato, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu D, Vemuri VK, Duclos RI Jr, Makriyannis A. The cannabinergic system as a target for anti-inflammatory therapies. Curr Top Med Chem. 2006;6(13):1401-26. doi: 10.2174/15680266106061401. PMID 16918457
- [Background] Moreira FA, Lutz B. The endocannabinoid system: emotion, learning and addiction. Addict Biol. 2008 Jun;13(2):196-212. doi: 10.1111/j.1369-1600.2008.00104.x. Epub 2008 Apr 16. PMID 18422832
- [Derived] Young TP, Erickson JS, Hattan SL, Guzy S, Hershkowitz F, Steward MD. A Single-Blind, Randomized, Placebo Controlled Study to Evaluate the Benefits and Safety of Endourage Targeted Wellness Formula C Sublingual +Drops in People with Post-Acute Coronavirus Disease 2019 Syndrome. Cannabis Cannabinoid Res. 2024 Feb;9(1):282-292. doi: 10.1089/can.2022.0135. Epub 2022 Oct 14. PMID 36252151
- See also: COVID-19 WHO — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: COVID-19 Infectious Disease Society of America (IDSA) — https://www.idsociety.org/practice-guideline/covid-19-guideline-treatment-and-management/